CLINICAL TRIAL: NCT05101538
Title: Anorexia Nervosa and it's Effects on Brain Function, Body Metabolism and Their Interaction
Brief Title: Anorexia Nervosa and Its Effects on Brain Function, Body Metabolism and Their Interaction
Acronym: AVAIN-PET
Status: Completed | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Principal Investigator, Pirjo Nuutila, Principal Investigator, Turku University Hospital
Other Study IDs: T113/2020
Record Dates: First submitted 2021-10-12; First posted 2021-11-01 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: Anorexia Nervosa
Keywords: Anorexia nervosa; metabolism; functional imaging; PET
MeSH Terms: conditions — Anorexia Nervosa

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients and controls: AN patients and controls are recruited, studied using imaging and followed for 5 years

SUMMARY:
The neuromolecular and metabolic underpinnings of Anorexia Nervosa (AN) are studied using multi-modal molecular (positron emission tomography with two different radioligands) and functional (functional magnetic resonance imaging) neuroimaging in a prospective design. Subjects with AN and normal weight adolescents will be studied with PET and MRI and followed for five years.

DETAILED DESCRIPTION:
A total of sixty females (30 with AN, 30 healthy controls) are recruited into this prospective study. The subjects will undergo physical examination, body tissue composition measurement, functional and structural MRI of the brain and body, and positron emission tomography (PET) with ligands [18F]-FDG, and [11C]carfentanil. Subjects' weight and physical condition will be followed up for 5 years. The study will start in August 2020 and end in the fall of 2028.

ELIGIBILITY:
Inclusion Criteria for AN:

1. Female sex
2. Age 18-32 3 years
3. BMI < 17.5 kg/m2
4. Currently fulfilling modified DSM-IV diagnosis of AN with or without amenorrhea, onset age before 25 years
5. Diagnosed less than 2 years ago

For controls:

1. Female sex
2. Age 18-32 3 years
3. BMI 19 20-25 kg/m2
4. No lifetime history of obesity (BMI ≥> 30) or eating disorders

Exclusion Criteria:

1. Any chronic disease or medication that could affect glucose metabolism or neurotransmission
2. History of psychiatric disorders (excl. AN for the corresponding study group)
3. Smoking of tobacco, taking of snuffs, or use of narcotics
4. Abusive use of alcohol

Ages: 18 Years to 32 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — AN is more frequent in females, rare in males.
Study Population: Totallly 30 female subjects with anorexia nervosa are recuited from the Eating Disorder Unit at the Turku University Hospital who meet the following criteria: i) modified DSM-IV diagnosis of AN with or without amenorrhea; ii) AN onset before the age of 25 years; iii) age between 18 and 32 3 years; iv) no lifetime history of binge eating. Their data are compared with 30 age and sex-matched healthy controls
Sampling Method: Probability Sample
Enrollment: 25 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2024-11-01 (Actual); Study Completion 2024-11-01 (Actual)

PRIMARY OUTCOMES:
Changes in brain reward system and metabolism in AN patients | 10 years
  AN patients and controls are studied using fMRI and PET imaging and followed 10 years. Reward system function is measured using functional MRI and metabolism using 18F-fluorodeoxy glucose and PETCT imaging
Predictive value of baseline body mass index (BMI), functional brain activation and metabolism in AN | 10 y
  Results from baseline are combined with follow updata

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD, PhD, Principal Investigator — Turku PET Centre, Turku University hospital
Locations (1):
- Turku PET Centre, Turku, Finland